CLINICAL TRIAL: NCT00043771
Title: Multi-Center, Double-Blind Study to Compare the Effects of 30mg Qd Versus 15 Mg Bid of Tolvaptan in Congestive Heart Failure Patients
Brief Title: Study to Compare the Effects of Two Dosages of Tolvaptan in Congestive Heart Failure Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 156-01-231
Record Dates: First submitted 2002-08-13; First posted 2002-08-14 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-09

CONDITIONS: Congestive Heart Failure
Keywords: CHF
MeSH Terms: conditions — Heart Failure | interventions — Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan

SUMMARY:
Patients with congestive heart failure will be assessed for safety and clinical effects of Tolvaptan 30 mg every day versus 15 mg twice a day over a period of 7 days.

ELIGIBILITY:
History of CHF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-05; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Central Cardiology Medical Clinic, Bakersfield, California
  - University of California-San Diego, San Diego, California
  - University of Miami/Jackson Memorial Hospital, Miami, Florida
  - Medical Research Institute, Slidell, Louisiana
  - Androscoggin Cardiology Associates, Auburn, Maine
  - University of Missouri-Kansas City School of Medicine, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Cardiology of Oklahoma, Tulsa, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina